CLINICAL TRIAL: NCT00173784
Title: Development of an Instrumental Activities of Daily Living Scale for Patients
Brief Title: Development of an Instrumental Activities of Daily Living Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361701231; NSC-94-2314-B-002-079
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Spinal Cord Injury
Keywords: psychometrics; activities of daily living
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This study is to develop an IADL Scale for patients with SCI (IADL-SCI) and examine its psychometric properties in three years.

DETAILED DESCRIPTION:
This study is to develop an IADL Scale for patients with SCI (IADL-SCI) and examine its psychometric properties in three years. In the first year, we will devote ourselves to the development of IADL-SCI - first version. About 150 patients will be recruited in this year.

In the second year, the study will be focused on investigating the psychometric properties of IADL-SCI in order to construct the formal version of IADL-SCI in about 120 patients with stable condition.

In the third year, we will be engaged in analyzing and comparing the psychometric properties of the three IADL scales (IADL-SCI, Frenchay Activities index, and Lawton IADL) to confirm that IADL-SCI is the best among the three. About 50 inpatients receiving rehabilitation will be recruited in this year.

ELIGIBILITY:
Inclusion Criteria:

patients with spinal cord injury

Exclusion Criteria:

patients with other major diseases (e.g., cancer)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-08; Study Completion 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: Jang Yuh, MPh, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University
Locations (1):
- School of Occupational Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan